CLINICAL TRIAL: NCT03173144
Title: Impact of Red and Processed Meat and Fibre Intake on Treatment Outcome Among Patients With Chronic Inflammatory Diseases: Protocol for a Prospective Cohort Study on Prognostic Factors and Personalised Medicine
Brief Title: Chronic Inflammatory Disease, Lifestyle and Treatment Response
Acronym: BELIEVE
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Hospital of Southern Jutland (Other); University Hospital Bispebjerg and Frederiksberg (Other); University of Copenhagen (Other); Odense University Hospital (Other); University of Aarhus (Other); Aalborg University Hospital (Other); Herning Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Sygehus Lillebaelt (Other); Aalborg University (Other); University of Kiel (Other); Colitis-Crohn Foreningen (Other); Herlev Hospital (Other); Regionshospitalet Silkeborg (Other); Aarhus University Hospital (Other); The Danish Psoriasis Association (Unknown)
Responsible Party: Principal Investigator, Vibeke Andersen, Professor, University of Southern Denmark
Other Study IDs: MOK1; 733100 (Other Grant/Funding Number: European Union's Horizon 2020 R.I.P.); KBF nr. 2016-056 (Other Grant/Funding Number: Odense Patient data Explorative Network); 2016-11-29 (Other Grant/Funding Number: Knud og Edith Eriksens Mindefond); J.nr 16/36626 (Other Grant/Funding Number: Region of Southern Denmark, University of Southern Denmark); OCAY-13-309 (Other Grant/Funding Number: Oak Foundation)
Record Dates: First submitted 2017-05-17; First posted 2017-06-01 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Autoimmune Diseases; Inflammatory Bowel Diseases; Crohn Disease (CD); Colitis, Ulcerative (UC); Arthritis, Rheumatoid (RA); Spondylarthropathies; Arthritis, Psoriatic (PsA); Psoriasis; Hidradenitis Suppurativa (HS); Uveitis
Keywords: Life Style; Diet; Food; Exercise; Treatment Outcome; Biomarkers; Smoking
MeSH Terms: conditions — Autoimmune Diseases; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Arthritis, Rheumatoid; Spondylarthropathies; Arthritis, Psoriatic; Psoriasis; Hidradenitis Suppurativa; Uveitis; Motor Activity; Smoking | interventions — Dietary Fiber

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Biospecimen Retention: Samples With DNA — blood, urine, feces, intestinal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Primary exposure variable — 1. Upper tertile (33.3% of the total sample) based on the ratio: fibre/meat intake is associated with better treatment outcome
  2. Low intake of red and processed meat (defined as below the lower tertile [33.3% of the total sample]) and high intake of dietary fibres (defined as those above the upper tertile [33.3% of the total sample]) are independently associated with better treatment outcome, and their synergy (interaction between the factors meat and fibres) gives the best treatment outcome
  Other Names: intake of red and processed meat and fibres
Other: Other (exploratory) exposure variables — * Lifestyle factors independently or combined (red and processed meat, vegetable, dietary fibre, cereals, gluten, legumes, red wine, dairy products, physical activity, smoking, total protein/ fat, protein/ fat from red and processed meat, glucemic index)
  * Pretreatment lifestyle-associated biomarkers
  * Combinations of lifestyle factors and lifestyle-associated biomarkers
  * Gene-environment interaction analyses
  * Pretreatment levels of inflammatory molecules

SUMMARY:
Chronic inflammatory diseases (CID) - including inflammatory bowel diseases (Crohn's disease and ulcerative colitis), rheumatic conditions (rheumatoid arthritis, axial spondyloarthritis, psoriatic arthritis), inflammatory skin diseases (psoriasis, hidradenitis suppurativa) and non-infectious uveitis are treated with biologics targeting the pro-inflammatory molecule tumour necrosis factor-α (TNF), i.e. TNF inhibitors. Up to one third of the patients do, however, not respond to biologics and lifestyle is assumed to affect the treatment outcome. However, little is known on the effects of lifestyle as a prognostic factor (possibly enabling personalised medicine). The aims of this multidisciplinary collaboration are to identify lifestyle factors that support individualised forecasting of optimised treatment outcome on these costly drugs.

This prospective cohort study will enrol CID patients assigned for biologic treatment. At baseline (Pre-treatment), patient characteristics are assessed using patient-reported outcome measures and clinical assessments on disease activity, quality of life, and lifestyle together with registry data on comorbidity and medication. Follow-up will be conducted at week 14-16 after treatment initiation (according to the current Danish standards). Evaluation of a successful treatment outcome response will - for each disease - be based on most frequently used primary endpoints; the major outcome of the analyses will be to detect differences in treatment outcome between patients with specific lifestyle characteristics.

The overarching goal of this project is to improve the lives of patients suffering from CID, by providing evidence to support dietary recommendations likely to improve the clinical outcome.

The study is approved by the local Ethics Committee (S-20160124) and the local Data Agency (2008-58-035). The study findings will be disseminated in peer-reviewed journals, via patient associations, and presented at national and international conferences.

DETAILED DESCRIPTION:
Chronic inflammatory diseases (CID), including inflammatory bowel diseases (IBD) (of which Crohn's disease [CD] and ulcerative colitis [UC] are the two most prevailed entities), rheumatic conditions (rheumatoid arthritis [RA], axial spondyloarthropathy [axSpA], psoriatic arthritis [PsA]), skin diseases (psoriasis [PsO], hidradenitis suppurativa [HS]), and eye disease (non-infectious uveitis [NiU]), are diseases of the immune system that are managed with biological agents targeting the pro-inflammatory cytokine tumour necrosis factor-α (TNF), i.e. TNF inhibitors.

Design In this prospective cohort study disease activity prior to and after (14-16 weeks) initiation of biologic treatment will be assessed. The endpoint is the treatment outcome defined as A: Responder according to the specific criteria described below (incl. drug-continuation) or B: Non-responder (incl. drug-discontinuation due to unacceptable side effects). Whether a patient will discontinue therapy is assumed to be based on a certain degree of shared decision making between the patient and physician supported by principles from national guidelines for each CID as recommended in the respective national guidelines and laboratory data.

Setting All patients assigned for initiation of biologic treatment at 1) Department of Gastroenterology and Hepatology, Aalborg University Hospital; 2) Department of Hepatology and Gastroenterology, Aarhus University Hospital; 3) Diagnostic Centre, Silkeborg Regional Hospital; 4) Department of Internal Medicine, Herning Regional Hospital; 5) Department of Gastroenterology, Herlev Hospital; 6) Organ Centre, Hospital of Southern Jutland; 7) Department of Gastroenterology Hospital of South West Jutland; 8) Department of Medical Gastroenterology, Department of Rheumatology, Department of Dermatology and Allergy Centre, and Department of Ophthalmology, Odense University Hospital from 1st of April 2017 and until 31th of Marts 2019 or until a minimum of 100 patients with IBD, 100 patients with RA, and 120 patients with axSpA, PsA, PsO, HS and NiU are achieved.

Clinical data consist of personal data, data on health and disease, lifestyle, laboratory measure, and disease activity scores including using patient-reported outcome measures (PROMs), clinical assessments, and laboratory data. Each participant will fill out validated questionnaires on disease activity, quality of life, and lifestyle using an electronic link. Studies have found electronic questionnaires to be equivalent to paper-based in relation to PROMs.

Data management The electronic questionnaire is in Danish language and the participants will have access to the questionnaire by an electronic link sent to their personal, electronic mailbox. All data will be stored in a secure research storage facility. Information registered by clinicians and technicians will be transferred from paper format to electronic format using either double entry of data or automated forms processing.

Statistical methods The investigators will use this rigorously designed, prospective cohort study to explore the ability to predict clinical response across the conditions included (Y=primary endpoint), and explore whether patients who are on a diet high in fibre AND low in red and processed meat (X=assessed at baseline) is an informative prognostic factor. Per default, the statistical model will include condition (any of the CID conditions included), and clinical centre (site #1 to #8) as fixed effects.

Sample size considerations: It is a well-known difficulty for exploratory prognostic factor research studies like this, to formalize how many participants (i.e. with events) to include. In order to consider an adequate number of outcome events, the investigators apply "the rule of thumb" that dictates that 10 outcome events are needed for each independent variable (possible predictors); the investigators plan to enrol 320 patients in total, and anticipate that 50% of these will experience a clinical response during the 14-16 week period after therapy is initiated. With this in mind: Anticipating that at least 160 will achieve clinical responses (among the 320 patients), this study will have a reasonable power to explore the impact of as many as 16 independent (predictor) variables (including condition and clinical centre).

Focusing on the contrast between groups, for a comparison of two independent binomial proportions (those with high fibre AND low meat intake vs other) using Pearson's Chi-square statistic with a Chi-square approximation with a two-sided significance level of 0.05 (P<0.05), a total sample size of 318 assuming an allocation ratio of 1 to 2 has an approximate power of 0.924 (i.e. >90% statistical power) when the proportions responding are 60% and 40%, respectively.

All the statistical programming will be done in SAS (Statistical Analysis Software), STATA or R, transparently reporting the source code used to analyse the data. All computational details will be available in the pre-specified Statistical Analysis Plan (will be finalised before data collection is complete).

Project organisation The project is organised with a Clinical Research Group and an Analytical Research Group. The clinical group includes specialists from the medical, gastroenterological, rheumatological, dermatological and ophthalmological departments that are sampling the cohort. The analytical group will perform the analyses on the biological material.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with chronic inflammatory disease
* initiation of targeted therapy
* able to read and understand Danish

Exclusion Criteria:

• not mentally able to reply the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: targeted therapy and able to read and understand Danish.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Clinical response to therapy depending on condition | week 14-16
  The predefined primary endpoint will be the proportion of patients with clinical response to therapy at first clinical follow-up.
  * Crohn's disease: HBI of 4 or less
  * Ulcerative colitis: Mayo Clinic Score of 2 or less (with no individual subscore of >1)
  * Rheumatoid arthritis: ACR20
  * Axial spondyloarthritis: ASAS20
  * Psoriatic arthritis: ACR20
  * Psoriasis: PASI75
  * Hidradenitis suppurativa: HiSCR
  * Uveitis: those who did not have a treatment failure

SECONDARY OUTCOMES:
Crohns disease: Disease-specific core outcome sets-1 | week 14-16
  • STRIDE (y/n)
Crohns disease: Disease-specific core outcome sets-2 | week 14-16
  • HBI (score)
Crohns disease: Disease-specific core outcome sets-3 | week 14-16
  • Physician global assessment (score)
Crohns disease: Disease-specific core outcome sets-4 | week 14-16
  • Number of draining fistulas (only fistulising CD) (number)
Crohns disease: Disease-specific core outcome sets-5 | week 14-16
  • Corticosteroid-Free Remission (y/n)
Crohns disease: Disease-specific core outcome sets-6 | week 14-16
  • Supplemental medication (y/n)
Ulcerative Colitis: Disease-specific core outcome sets-1 | week 14-16
  • STRIDE criteria (y/n)
Ulcerative Colitis: Disease-specific core outcome sets-2 | week 14-16
  • Mayo Clinical Score (score)
Ulcerative Colitis: Disease-specific core outcome sets-3 | week 14-16
  • Mayo "normal mucosal appearance" (y/n)
Ulcerative Colitis: Disease-specific core outcome sets-4 | week 14-16
  • Mayo clinical response (y/n)
Ulcerative Colitis: Disease-specific core outcome sets-5 | week 14-16
  • SCCAI (score)
Ulcerative Colitis: Disease-specific core outcome sets-6 | week 14-16
  • Corticosteroid-Free Remission (y/n)
Ulcerative Colitis: Disease-specific core outcome sets-7 | week 14-16
  • Supplemental medication (y/n)
Rheumatoid Arthritis: Disease-specific core outcome sets-1 | week 14-16
  • Tender joints (number)
Rheumatoid Arthritis: Disease-specific core outcome sets-2 | week 14-16
  • Swollen joints (number)
Rheumatoid Arthritis: Disease-specific core outcome sets-3 | week 14-16
  • Pain (0-100 mm VAS)
Rheumatoid Arthritis: Disease-specific core outcome sets-4 | week 14-16
  • Physician global assessment (0-100 mm VAS)
Rheumatoid Arthritis: Disease-specific core outcome sets-5 | week 14-16
  • Patient global assessment (0-100 mm VAS)
Rheumatoid Arthritis: Disease-specific core outcome sets-6 | week 14-16
  • HAQ-DI (score)
Rheumatoid Arthritis: Disease-specific core outcome sets-7 | week 14-16
  • C-Reactive protein (mg/l)
Rheumatoid Arthritis: Disease-specific core outcome sets-8 | week 14-16
  • DAS28-CRP (score)
Rheumatoid Arthritis: Disease-specific core outcome sets-9 | week 14-16
  • Simplified Disease Activity Index (SDAI) (index)
Axial Spondyloarthropathy: Disease-specific core outcome sets-1 | week 14-16
  • BASFI (score)
Axial Spondyloarthropathy: Disease-specific core outcome sets-2 | week 14-16
  • BASDAI (score)
Axial Spondyloarthropathy: Disease-specific core outcome sets-3 | week 14-16
  • BASMI (score)
Axial Spondyloarthropathy: Disease-specific core outcome sets-4 | week 14-16
  • Total score for back pain (0-100 mm VAS)
Axial Spondyloarthropathy: Disease-specific core outcome sets-5 | week 14-16
  • Physician global assessment (0-100 mm VAS)
Axial Spondyloarthropathy: Disease-specific core outcome sets-6 | week 14-16
  • Patient global assessment (0-100 mm VAS)
Axial Spondyloarthropathy: Disease-specific core outcome sets-7 | week 14-16
  • C-Reactive protein (mg/l)
Psoriatic Arthritis: Disease-specific core outcome sets-1 | week 14-16
  • Tender joints (number)
Psoriatic Arthritis: Disease-specific core outcome sets-2 | week 14-16
  • Swollen joints (number)
Psoriatic Arthritis: Disease-specific core outcome sets-3 | week 14-16
  • Psoriatic Arthritis Pain VAS (0-100 mm VAS)
Psoriatic Arthritis: Disease-specific core outcome sets-4 | week 14-16
  • Physician global assessment (0-100 mm VAS)
Psoriatic Arthritis: Disease-specific core outcome sets-5 | week 14-16
  • Patient global assessment (0-100 mm VAS)
Psoriatic Arthritis: Disease-specific core outcome sets-6 | week 14-16
  • HAQ-DI (score)
Psoriatic Arthritis: Disease-specific core outcome sets-7 | week 14-16
  • C-Reactive protein (mg/l)
Psoriatic Arthritis: Disease-specific core outcome sets-8 | week 14-16
  • DAS28-CRP (score)
Psoriatic Arthritis: Disease-specific core outcome sets-9 | week 14-16
  • Simplified Disease Activity Index (SDAI)(score)
Psoriatic Arthritis: Disease-specific core outcome sets-10 | week 14-16
  • PASI (score)
Psoriasis: Disease-specific core outcome sets-1 | week 14-16
  • PASI (score)
Psoriasis: Disease-specific core outcome sets-2 | week 14-16
  • Physician global assessment (0-100 mm VAS)
Psoriasis: Disease-specific core outcome sets-3 | week 14-16
  • Patient global assessment (0-100 mm VAS)
Psoriasis: Disease-specific core outcome sets-4 | week 14-16
  • Dermatology Life Quality Index (DLQI) Total Score (score)
Hidradenitis Suppurativa: Disease-specific core outcome sets-1 | week 14-16
  • Participants who achieve Abscess and Inflammatory Nodule (AN) Count of 0, 1, and 2, respectively (score)
Hidradenitis Suppurativa: Disease-specific core outcome sets-2 | week 14-16
  • Patient's Global Assessment of Skin Pain (0-100 mm VAS)
Hidradenitis Suppurativa: Disease-specific core outcome sets-3 | week 14-16
  • Modified Sartorius Score (score)
Non-Infectious Uveitis: Disease-specific core outcome sets-1 | week 14-16
  • New active, inflammatory chorioretinal or retinal vascular lesions relative to Baseline (y/n)
Non-Infectious Uveitis: Disease-specific core outcome sets-2 | week 14-16
  • Inability to achieve ≤ 0.5+ or a 2-step increase relative to best state achieved at all visits in anterior chamber cell grade or vitreous haze grade (y/n)
Non-Infectious Uveitis: Disease-specific core outcome sets-3 | week 14-16
  • Worsening of best corrected visual acuity by ≥ 15 letters relative to best state achieved (y/n)
Health-related quality of life-1 | week 14-16
  • SF12 (Short Form Health Survey) (score)
Health-related quality of life and disability-2 | week 14-16
  • SHS (Short Health Scale) (score)
Health-related quality of life-2 | week 14-16
  • SHS (Short Health Scale) (score)
Global assessment-1 | week 14-16
  • Physician global assessment (0-100 mm VAS)
Global assessment-2 | week 14-16
  • Patient global assessment (0-100 mm VAS)

OTHER OUTCOMES:
Exploratory outcome measure - Serious adverse events | week 14-16
  • Serious adverse events (y/n)
Biological response | week 14-16
  • CRP (mg/l)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Andersen, Prof, Principal Investigator — University of Southern Denmark
Locations (3):
- Denmark (3):
  - Hospital of Southern Jutland, Aabenraa
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Pseudoanonymised data on Health, lifestyle, treatment response and biological analyses will be shared with the Horizon 2020-project "A Systems medicine approach to chronic inflammatory disease" (SYSCID) partners.

REFERENCES:
- [Derived] Eggers KR, Mollegaard KM, Gregersen L, Overgaard SH, Hikmat Z, Ellingsen T, Kjeldsen J, Pedersen AK, Petersen SR, Jawhara M, Nexoe AB, Bygum A, Hvas CL, Dahlerup JF, Bergenheim FO, Glerup H, Brodersen JB, Munk HL, Pedersen N, Nielsen OH, Andersen KW, Heitmann BL, Christensen R, Andersen V. Impact of Obesity on Treatment Response in Patients With Chronic Inflammatory Disease Receiving Biologic Therapy: Secondary Analysis of the Prospective Multicentre BELIEVE Cohort Study. Scand J Immunol. 2025 Jun;101(6):e70035. doi: 10.1111/sji.70035. PMID 40545788
- [Derived] Larsen MGR, Overgaard SH, Petersen SR, Mollegaard KM, Munk HL, Nexoe AB, Glerup H, Guldmann T, Pedersen N, Saboori S, Dahlerup JF, Hvas CL, Andersen KW, Jawhara M, Haagen Nielsen O, Bergenheim FO, Brodersen JB, Bygum A, Ellingsen T, Kjeldsen J, Christensen R, Andersen V. Effects of smoking on clinical treatment outcomes amongst patients with chronic inflammatory diseases initiating biologics: secondary analyses of the prospective BELIEVE cohort study. Scand J Immunol. 2024 Sep;100(3):e13395. doi: 10.1111/sji.13395. Epub 2024 Jul 7. PMID 38973149
- [Derived] Overgaard SH, Sorensen SB, Munk HL, Nexoe AB, Glerup H, Henriksen RH, Guldmann T, Pedersen N, Saboori S, Hvid L, Dahlerup JF, Hvas CL, Jawhara M, Andersen KW, Pedersen AK, Nielsen OH, Bergenheim F, Brodersen JB, Heitmann BL, Halldorsson TI, Holmskov U, Bygum A, Christensen R, Kjeldsen J, Ellingsen T, Andersen V. Impact of fibre and red/processed meat intake on treatment outcomes among patients with chronic inflammatory diseases initiating biological therapy: A prospective cohort study. Front Nutr. 2022 Oct 13;9:985732. doi: 10.3389/fnut.2022.985732. eCollection 2022. PMID 36313095
- [Derived] Christensen R, Heitmann BL, Andersen KW, Nielsen OH, Sorensen SB, Jawhara M, Bygum A, Hvid L, Grauslund J, Wied J, Glerup H, Fredberg U, Villadsen JA, Kjaer SG, Fallingborg J, Moghadd SAGR, Knudsen T, Brodersen J, Frojk J, Dahlerup JF, Bojesen AB, Sorensen GL, Thiel S, Faergeman NJ, Brandslund I, Bennike TB, Stensballe A, Schmidt EB, Franke A, Ellinghaus D, Rosenstiel P, Raes J, Boye M, Werner L, Nielsen CL, Munk HL, Nexoe AB, Ellingsen T, Holmskov U, Kjeldsen J, Andersen V. Impact of red and processed meat and fibre intake on treatment outcomes among patients with chronic inflammatory diseases: protocol for a prospective cohort study of prognostic factors and personalised medicine. BMJ Open. 2018 Feb 8;8(2):e018166. doi: 10.1136/bmjopen-2017-018166. PMID 29439003